CLINICAL TRIAL: NCT03679923
Title: Efficacy of NEM® Brand Eggshell Membrane Versus Placebo in Exercised-induced Joint Pain, Stiffness, & Cartilage Turnover in Healthy Men & Women
Brief Title: NEM® Versus Placebo in Exercised-induced Joint Pain, Stiffness, & Cartilage Turnover in Healthy Men & Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Collaborators: QPS Bio-Kinetic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ESM-CLN#2018T02
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Exercise-induced Joint Pain; Exercise-induced Joint Stiffness; Exercise-induced Joint Cartilage Turnover
Keywords: exercise-induced; joint pain; joint stiffness; cartilage turnover; CTX-II
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Intervention Model Description: treatment versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEM® brand eggshell membrane (Experimental): NEM, 500 mg, #0 capsule, once daily orally for 2 weeks
  Interventions: Dietary Supplement: NEM® brand eggshell membrane
- Placebo (Placebo Comparator): Placebo, 500 mg, #0 capsule, once daily orally for 2 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NEM® brand eggshell membrane — Dietary supplement for the support of joint health.
  Other Names: Natural Eggshell Membrane
  Arms: NEM® brand eggshell membrane
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is intended to evaluate the effect of the dietary supplement NEM® brand eggshell membrane versus placebo in reducing exercise-induced joint pain, stiffness & cartilage turnover in healthy men & women. Half of the study participants will receive NEM, once daily, orally while the other half of the study participants will receive placebo, once daily, orally while performing an exercise regimen every other day for two weeks.

DETAILED DESCRIPTION:
Moderate exercise can induce discomfort in joints when done infrequently or when done too intensely or for too long a period. This discomfort is often realized as either pain or stiffness in the joint that was the focus of the exercise. For example, one's knees will hurt after jogging for several miles, particularly if jogging for the first time. This study is intended to evaluate whether NEM® brand eggshell membrane can alleviate joint pain or stiffness, either directly following exercise or 12 hours post-exercise versus placebo. The study will also evaluate NEM's effect, on cartilage turnover via the cartilage degradation biomarker c-terminal cross-linked telopeptide of type II collagen (CTX-II). Participants will perform a minimum of 40 steps per leg utilizing an aerobics step at the clinical site. They will follow this exercise regimen on alternating days for 2 consecutive weeks. Changes in pain & stiffness (immediate & 12-hour) will be compared to both baseline and to the placebo group. Urine samples will also be collected at baseline and at the end of Week 1 & Week 2. The change in CTX-II from baseline will be compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects must be 40-75 years of age at the time of Screening.
2. Subjects must not have been diagnosed with a JCT disease (i.e. osteoarthritis, rheumatoid arthritis, spondyloarthritis, bursitis, gout, systemic lupus erythematosus, fibromyalgia, etc.) affecting the hip, knee, or ankle by a licensed physician prior to enrollment evaluation / screening.
3. Subjects must have a resting pain/discomfort score of ≤ 2 on the 10-point continuous scale in the knee with the most severe pain/discomfort at the Follow-Up Screening/Baseline (first exercise visit).
4. Subjects must be willing and healthy enough, as judged by the clinical Investigator or Sub-Investigator(s), to perform moderate exercise.
5. Subjects must be available for and willing to attend all evaluation visits.
6. Subjects must be able and willing to give informed consent.
7. Subjects must be willing to use only acetaminophen as rescue pain medication, if needed.
8. Subjects participating in prior studies evaluating eggshell membrane, curcumin, fish oil or collagen can participate in the present study so long as they are not currently taking an eggshell membrane, fish oil, curcumin, or collagen supplement and have not done so for 60 days prior to screening.

Exclusion Criteria:

1. Subject is currently receiving therapy with remission-inducing drugs (i.e. methotrexate, TNF biologics, etc.), immunosuppressive drugs (i.e. corticosteroids, transplantation medications, etc.) or planning to use these products during the study period.
2. Subject has been diagnosed with any clinically significant confounding inflammatory disease or condition that would interfere with the study evaluation, as judged by the clinical investigator (i.e. pseudo gout, Paget's disease, chronic pain syndrome, active rheumatic fever, etc.).
3. Subject has known allergy to any of the investigational products, including but not limited to eggs or egg products and rice or rice flour. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study.
4. Subject suffers from clinically significant cardiac, pulmonary, or other complications that would prevent them from performing moderate exercise or could pose a risk to the subject's health, as judged by the clinical investigator.
5. Subject participates in activities involving intensive use of the lower extremities (i.e. running / jogging, sports, bicycling, dancing, etc.) 2 or more days per week or participates in activities that involve moderate use of the lower extremities (i.e. walking, golfing, yoga, etc.) 3 or more days per week.
6. Subject's body weight is greater than 300 pounds (136.1 kg) at the time of Screening.
7. Subject is currently taking or is unwilling to forgo the use of prescription, over-the-counter (OTC) treatments, and/or dietary supplements affecting joint health within 30 days prior to baseline evaluation and for the duration of the study. Prohibited medications include: NSAIDs, analgesics (other than acetaminophen), opioids, anti-depressants (of all drug classes for this indication, including but not limited to SSRI's such as citalopram and fluoxetine, TCA's such as amitriptyline and amoxapine, SNRI's such as duloxetine or SNRI's used for fibromyalgia such as milnacipran and NDRI's such as bupropion), other medications for the management of painful conditions (i.e. fibromyalgia) including gabapentin and tizanidine & joint supplements. Examples of these types of medications are: aspirin, ibuprofen, naproxen, oxycodone, propoxyphene, diclofenac, celecoxib, amitriptyline, duloxetine, glucosamine, chondroitin, MSM, white willow bark, turmeric or curcumin, Boswellia, fish oil, etc.

   a. Washout Periods: Subjects are eligible to participate in the study following a 7-day washout period for opioids, a 14-day washout period for analgesics & NSAIDs, and a 90-day washout period for steroids, anti-depressants, or JCT dietary supplements (i.e. glucosamine, chondroitin, MSM, etc.) Acetaminophen must not have been taken within 24 hours of the first baseline evaluation.
8. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of the first baseline evaluation.
9. Pregnant and breastfeeding women, or women who intend to become pregnant during the course of the study.
10. Subject has a history or positive test result of HIV, hepatitis B or hepatitis C.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Exercise-induced Cartilage Turnover via CTX-II Biomarker | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced cartilage turnover in healthy men & women by evaluating the change in urinary CTX-II levels.

SECONDARY OUTCOMES:
Exercise-induced Joint Pain via questionnaire | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced knee discomfort (pain/aching) based upon perceived pain rated on a 0-10 point continuous scale (where 0 = no pain)..
Exercise-induced Joint Stiffness via questionnaire | 2 weeks
  To evaluate the efficacy of NEM® versus placebo at reducing exercise-induced knee stiffness based upon perceived stiffness rated on a 0-10 point continuous scale (where 0 = no stiffness).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ruff, Ph.D., Study Chair — ESM Technologies, LLC; Christopher Bailey, Ph.D., Study Director — ESM Technologies, LLC; Kayce Morton, D.O., Principal Investigator — QPS Bio-Kinetic
Locations (1):
- QPS Bio-Kinetic, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruff KJ, Morton KM, Duncan SA, Back M. Eggshell Membrane (NEM®) Reduces Exercise-Induced Joint Pain, Stiffness and Cartilage Turnover in Healthy Men and Women: A Randomized Controlled Trial. Int J Phys Med Rehabil. (2024) 12:722.
- See also: International Journal of Physical Medicine & Rehabilitation Website — https://www.longdom.org/open-access/eggshell-membrane-nem-reduces-exerciseinduced-joint-pain-stiffness-and-cartilage-turnover-in-healthy-men-and-women-a-randomized-co-106640.html